CLINICAL TRIAL: NCT04455269
Title: The Efficacy of Full Mouth Erythritol Powder Air-Polishing Therapy (FM-EPAPT) Versus Traditional Ultrasonic Debridment (UD): a Randomized Controlled Study.
Acronym: ERICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Magda Mensi, principal investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERICO np: 2637
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Gingivitis
Keywords: Gingivitis; GBT; Ultrasonic debridement
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Mono-centric, double-blinded, randomized clinical trial (RCT) with a split-mouth design.
Who Masked: Investigator
Masking Description: Clinical examination, collection of periodontal parameters and clinical photographs were performed by the same trained dentist blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full-Mouth Erythritol Powder Air-polishing Therapy (FM-EPAPT) (Experimental): The quadrants allocated to FM-EPAPT underwent the following steps:
  * Decontamination of soft tissues with air-polishing and erythritol powder;
  * Supra-gingival removal biofilm with air-polishing and erythritol powder;
  * Sub-gingival removal of biofilm with air-polishing and erythritol;
  * Calculus removal with a piezoceramic scaler.
  Interventions: Device: AIRFLOW® with PLUS® powder and PIEZON® scaler
- Ultrasonic debridement and abrasive paste (US+P) (Active Comparator): The quadrants allocated to US+P treatment underwent the following steps:
  * Full-mouth ultrasonic debridement with piezoceramic scaler;
  * Plaque removal and polishing with soft rubber cup and low-RDA polishing paste
  Interventions: Device: PIEZON® scaler and rubber cup with abrasive paste

INTERVENTIONS:
Device: AIRFLOW® with PLUS® powder and PIEZON® scaler — Air-polishing will be use as main instrument for biofilm and stains removal, followed by ultrasonic scaling
  Arms: Full-Mouth Erythritol Powder Air-polishing Therapy (FM-EPAPT)
Device: PIEZON® scaler and rubber cup with abrasive paste — Application of ultrasonic scaler on the entire dentition, followed by residual biofilm and stains removal and polishing
  Arms: Ultrasonic debridement and abrasive paste (US+P)

SUMMARY:
Traditional methods for plaque and calculus removal involve the use of mechanical and/or manual instruments, followed by surface polishing with rubber cups and low abrasive pastes. These instruments may cause the unintended removal of hard dental tissue, such as enamel, cementum and dentine, increasing surface roughness. Moreover, they can lead to gingival recession and consequent hypersensitivity and discomfort during treatment. New minimally-invasive approaches to biofilm removal have been recently introduced with the aim to limit the negative impact on the oral tissue. Air-polishing with low-abrasiveness powders are proven suitable for both for supra- and sub-gingival plaque removal. The use of low-abrasiveness powders could lead to several advantages, such as reduction of treatment discomfort, shorter treatment time, the possibility of cleaning areas with difficult access and minor damage on soft and hard tissues.

Aim: the aim of this study is to evaluate the efficacy of the Full Mouth Erithrytol Powder Air-Polishing Therapy compared to traditional ultrasonic debridment (UD) and polishing in patient affected by gingivitis.

Test hypotesis: there is no difference in clinical outcome between two methods against the hypothesis of a difference in terms of changes in Blending on Probing (BOP).

To test this hypothesis, the patients, upon initial evaluation, were treated in split mouth:

* The control group undergoing the standard procedure with full-mouth ultrasonic debridement and polishing with rubber cup and abrasive paste.
* The study group undergoing an innovative procedure involving full-mouth air-polishing followed by ultrasonic calculus removal.

Follow-ups are scheduled at 2 weeks and 1, 3, 6 and 12 months.

DETAILED DESCRIPTION:
TRIAL DESIGN:

Mono-centric, pragmatic, double-blinded, randomized clinical trial (RCT) with split-mouth design. The trial will have a one year of duration.

PRIMARY OUTCOME:

- Change in BoP: change in percentage of sites positive to bleeding on probing.

SECONDARY OUTCOMES:

* Change in Plaque Index (PI): change in percentage of sites with presence of plaque. Baseline values will be compared to the values recorded at follow-up visits.
* Change in Residual Plaque Area (RPA): Post-treatment percentage of tooth area with residual plaque, visualised via plaque disclosing agent. This will be calculated with computer software analysis (ImageJ) on clinical photographs.
* Change in Periodontal Attachment Level (PAL): change in mean value for each patient will be calculated. Baseline values will be compared to the values recorded at follow-up visits.
* Change in (Pocket Probing Depth) PPD: change in mean value for each patient will be calculated. Baseline values will be compared to the values recorded at follow-up visits.
* Duration of the treatment: calculated in minutes. Time will be recorded starting from the opening the randomisation envelope until the clinician is satisfied with the clinical result.
* Comfort of the patient: an anonymous questionnaire will be administered at baseline and each recall appointment.
* Sensation of cleanliness: an anonymous questionnaire will be administered at baseline and each recall appointment.

STUDY POPULATION:

41 Systemically healthy patients affected by gingivitis will be included in this study. Presence of gingivitis is defined as: absence of Probing pocket depth (PPD) > 4mm and presence of BoP >25%.

INCLUSION CRITERIA:

* Patients affected by gingivitis (BoP >25%);
* Patients with at least 5 teeth per quadrant;
* Systemically healthy;
* Age > 18 years;
* Smoking less than 10 cigarettes a day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gingivitis (BoP > 25%);
* Presence of at least 5 teeth per quadrant;
* Systemically healthy;
* Age between 20 and 40 years old.

Exclusion Criteria:

* Presence of periodontal disease, defined as >3 mm of clinical attachment loss at any site;
* Presence of fixed retainers, orthodontic appliances or complex prothetic restorations;
* Presence of crowding;
* Pregnant or lactating;
* Allergy to chlorhexidine or erythritol;
* Smoking >10 cigarettes per day;
* Unwillingness to undergo the proposed treatment and recalls;

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Bleeding on Probing (BoP) | study completion, an average of 18 months
  Change in percentage of sites positive to bleeding on probing

SECONDARY OUTCOMES:
Change in Plaque Index (PI) | From baseline to study completion (12 months)
  Change in percentage of site with plaque. Baseline values will be compared to the values recorded in the follow-up visits.
Change in residual plaque area (RPA) | From baseline to study completion (12 months)
  Post-treatment residual plaque recorded via plaque disclosing agent, clinical photographs and image software analysis
Change in Periodontal Attachment Level (PAL) | From baseline to study completion (12 months)
  Change in mean PAL value for each patient should be calculated. Baseline values will be compared to the values recorded in the follow-up visits.
Change in Pocket Probing Depth (PPD) | From baseline to study completion (12 months)
  Change in mean PPD value for each patient. Baseline values will be compared to the values recorded in the follow-up visits.
Treatment time | From baseline to study completion (12 months)
  Calculated in minutes, from the opening of the randomisation envelope to the end of the instrumentation.
Comfort of the patient | From baseline to study completion (12 months)
  An anonymous questionnaire will be administered at baseline and each recall appointment. The score is on a scale: from 0 to 5, where 0 is the minimum discomfort and 5 the maximum discomfort.
Sensation of cleanliness | From baseline to study completion (12 months)
  An anonymous questionnaire will be administered at baseline and each recall appointment. The score is on a scale of 5 feelings: insufficient, sufficient, average, good and optimal.

CONTACTS AND LOCATIONS:
Overall Officials: Magda Mensi, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- Magda Mensi, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Draenert ME, Jakob M, Kunzelmann KH, Hickel R. The prevalence of tooth hypersensitivity following periodontal therapy with special reference to root scaling. A systematic review of the literature. Am J Dent. 2013 Feb;26(1):21-7. PMID 23724545
- [Result] Buhler J, Amato M, Weiger R, Walter C. A systematic review on the patient perception of periodontal treatment using air polishing devices. Int J Dent Hyg. 2016 Feb;14(1):4-14. doi: 10.1111/idh.12119. Epub 2015 Jan 23. PMID 25619863
- [Result] Flemmig TF, Arushanov D, Daubert D, Rothen M, Mueller G, Leroux BG. Randomized controlled trial assessing efficacy and safety of glycine powder air polishing in moderate-to-deep periodontal pockets. J Periodontol. 2012 Apr;83(4):444-52. doi: 10.1902/jop.2011.110367. Epub 2011 Aug 23. PMID 21861637
- [Result] Camboni S, Donnet M. Tooth Surface Comparison after Air Polishing and Rubber Cup: A Scanning Electron Microscopy Study. J Clin Dent. 2016 Mar;27(1):13-18. PMID 28390211
- [Result] Kim SY, Kang MK, Kang SM, Kim HE. Effects of ultrasonic instrumentation on enamel surfaces with various defects. Int J Dent Hyg. 2018 May;16(2):219-224. doi: 10.1111/idh.12339. Epub 2018 Mar 13. PMID 29532597